CLINICAL TRIAL: NCT05113797
Title: Use of the OPTIMAL Theory of Motor Learning With the Lower Quarter Y-Balance Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Darren Q. Calley, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-009316
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Subjects will perform YBT-LQ practice tests using standardized set of verbal instructions provided in the YBT-LQ online manual prior to the testing condition.
  Interventions: Diagnostic Test: Lower Quarter Y-Balance Test
- OPTIMAL Motor Learning Group (Experimental): Subjects will perform the YBT-LQ with the practice period altered to implement aspects of the three pillars of the OPTIMAL motor learning theory (promotion of autonomy support (AS), presence of an external focus (EF) of attention, and implementation of enhanced expectancies (EE) placed upon a task).
  Interventions: Diagnostic Test: Lower Quarter Y-Balance Test; Behavioral: OPTIMAL motor learning theory

INTERVENTIONS:
Diagnostic Test: Lower Quarter Y-Balance Test — Dynamic balance assessment performed in a standing position while balanced on one leg, participants are asked to move a plastic box with their other foot in three directions (forward, back to the left, and back to the right) and a distance measurement is recorded. Each leg will be tested three times in each direction for the YBT-LQ assessment.
Behavioral: OPTIMAL motor learning theory — OPTIMAL theoretical framework instructions and coaching will be utilized to improve motor performance through three main components: promotion of autonomy support (AS), presence of an external focus (EF) of attention, and implementation of enhanced expectancies (EE) placed upon a task.
  Arms: OPTIMAL Motor Learning Group

SUMMARY:
Assessing and improving movement quality are important components of rehabilitation. The Lower Quarter Y-Balance Test (YBT-LQ) is a balance test used to assess dynamic balance in healthy adults, athletes, and those who are rehabilitating a lower extremity injury. Performing the YBT-LQ requires utilization of different strategies. It is unknown how different practice conditions will affect dynamic balance learning or performance on YBT-LQ. This study aims to compare the influence of OPTIMAL motor learning practice with standard practice conditions on YBT-LQ measurements.

DETAILED DESCRIPTION:
The Lower Quarter Y-Balance Test (YBT-LQ) is used to assess dynamic balance and functional symmetry in healthy adults, athletes, and those who are rehabilitating a lower extremity injury, and has good to excellent interrater reliability. Performing the YBT-LQ requires utilization of different neuromotor and postural control strategies in each direction of the test. The OPTIMAL theory of motor learning is a theoretical framework that has been shown to improve motor performance through three main components: promotion of autonomy support (AS), presence of an external focus (EF) of attention, and implementation of enhanced expectancies (EE) placed upon a task. These components of the OPTIMAL theory of motor learning have been demonstrated to enhance balance learning in several populations. There is also extensive literature on the effects of the individual components of the OPTIMAL theory of motor learning and some evidence that demonstrates the beneficial effects of the combined components on motor learning. However, to the authors knowledge, literature has not been published upon the effect of all three components of the OPTIMAL theory of motor learning on dynamic balance learning. Therefore, the purpose of this study is intended to determine if the OPTIMAL theory of motor learning will influence performance on the YBT-LQ.

Healthy participants aged 18 to 65 will be recruited for participation through word-of-mouth advertising. Inclusion criteria will include a passing score of >35 degrees bilateral ankle dorsiflexion and an ability to balance on one leg. Upon signing the informed consent document from participants, height, weight, BMI, gender, age, and limb length will be recorded for data analysis. Participants will be randomly assigned to one of two groups: an OPTIMAL motor learning group or a control group. The intended experimental design will be a multigroup nonequivalent pretest-posttest control group for this study. Participants will attend two study visits separated by 2-14 days. A visit one baseline YBT-LQ pretest will be administered in a standardized fashion the same for both groups. During visit two, the OPTIMAL group will practice the YBT-LQ using OPTIMAL principles, while the control group practices the YBT-LQ using standard principles, then both groups will undergo a posttest YBT-LQ measurement. Primary outcome measures will be normalized composite scores of the YBT-LQ. Secondary outcome measures will be participant self-reported measures of perceived competence, task effort, level of autonomy, and externally focused attention during the task on a 0 to 10 Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Having the ability to safely stand on one leg and pass the ankle dorsiflexion clearing test (> 35 degrees ankle dorsiflexion).

Exclusion Criteria:

* Presence of a recent lower extremity injury in the last month that limits their ability to stand on one leg.
* Failure to achieve 35 degrees of bilateral dorsiflexion on the dorsiflexion clearing test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change in composite YBT-LQ scores | Baseline, 14 days
  Measure by 3 reach trials in 3 directions on each leg recorded to the nearest 0.5 cm. Composite score calculated by the sum of three directions for one leg divided by three times limb length, multiplied by 100

SECONDARY OUTCOMES:
Perceived competence | 14 days
  Measured using a self-reported Likert scale that rates their level of agreement to the statement, "I had the ability and understanding to move the box as far as possible in all three directions (anterior, posteromedial, and posterolateral)" on a scale of 0=strongly disagree, 5=neutral, and 10=strongly agree
Task Effort | 14 days
  Measured using a self-reported Likert scale that rates their level of agreement to the statement, "I tried very hard on this balance test" on a scale of 0=strongly disagree, 5=neutral, and 10=strongly agree
Level of autonomy | 14 days
  Measured using a self-reported Likert scale that rates their level of agreement to the statement, "I felt in control of my ability to perform well on the Lower Quarter Y-Balance Test" on a scale of 0=strongly disagree, 5=neutral, and 10=strongly agree
Externally focused attention during the task | 14 days
  Measured using a self-reported Likert scale that rates their level of agreement to the statement, "I focused on the target more than myself pushing the box during the test" on a scale of 0=strongly disagree, 5=neutral, and 10=strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Darren Calley, PT, DScPT, OCS, Principal Investigator — Mayo Clinic
Locations (1):
- Darren Calley, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials